CLINICAL TRIAL: NCT01553019
Title: A Phase II Trial of Postoperative Proton Radiotherapy With Concomitant Chemotherapy for Patients With Resected Pancreatic Adenocarcinoma
Brief Title: Postoperative Proton Radiotherapy With Chemo for Pancreatic Cancer
Acronym: PC03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 1013-PC03
Record Dates: First submitted 2011-10-21; First posted 2012-03-13 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Pancreatic Cancer
Keywords: Proton radiation; Chemotherapy; Pancreatic cancer; Postoperative
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Proton Therapy; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1- R(0) negative (Experimental): 50.40 cobalt gray equivalent (CGE) Proton Radiation and concomitant chemotherapy with weekly gemcitabine
  Interventions: Radiation: Proton radiation; Drug: Gemcitabine
- 2- R(1) micro-positive (Experimental): 54.00 cobalt gray equivalent(CGE) Proton Radiation and concomitant chemotherapy with weekly gemcitabine
  Interventions: Radiation: Proton radiation; Drug: Gemcitabine
- 3- R(2) gross positive (Experimental): 59.40 cobalt gray equivalent (CGE) Proton Radiation and concomitant chemotherapy with weekly gemcitabine
  Interventions: Radiation: Proton radiation; Drug: Gemcitabine

INTERVENTIONS:
Radiation: Proton radiation — Proton Radiation Therapy: R(0) negative ... 50.40 cobalt gray equivalent (CGE) at 1.8 CGE per fraction ; R(1) micro-positive ...54.00 CGE at 1.8 CGE per fraction; R(2) gross positive...59.40 CGE at 1.8 CGE per fraction
Drug: Gemcitabine — Gemcitabine 300 mg/m2 infused over 30 minutes, weekly during proton therapy.
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, proton radiation combined with chemotherapy has on resected pancreatic cancer.

DETAILED DESCRIPTION:
Proton radiation with concomitant chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of primary head of pancreas invasive adenocarcinoma managed with a potentially curative resection
* Post resection CA19-9 tumor marker baseline

Exclusion Criteria:

- Previous history of invasive malignancy (except non-melanoma skin cancer and low to intermediate risk prostate cancer) unless the patient has been disease free for at least 5 years prior to study consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-10; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Radiation Toxicity | 90 days after completion of RT
  Assessment of acute/late severe (defined as grade 3-5) radiation toxicity at the completion of therapy. Acute toxicity will be defined to be toxicity occurring within 90 days from the start of radiation treatment, and late toxicity will be defined as toxicity occurring more than 90 days from the start of radiation treatment.

SECONDARY OUTCOMES:
Survival Rate | 1 year after completion of RT
  One year overall survival rate
Response rate via CA 19-9 | Every 3 months for 2 years, then every 6 months for 3-5 years then annually thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Romaine C Nichols, MD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (2):
- United States (2):
  - University of Florida Proton Therapy Institute, Jacksonville, Florida
  - Provision Proton Therapy Center, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tepper J, Nardi G, Sutt H. Carcinoma of the pancreas: review of MGH experience from 1963 to 1973. Analysis of surgical failure and implications for radiation therapy. Cancer. 1976 Mar;37(3):1519-24. doi: 10.1002/1097-0142(197603)37:33.0.co;2-o. PMID 1260670
- [Background] Gudjonsson B. Cancer of the pancreas. 50 years of surgery. Cancer. 1987 Nov 1;60(9):2284-303. doi: 10.1002/1097-0142(19871101)60:93.0.co;2-v. PMID 3326653
- [Background] Regine WF, Winter KA, Abrams RA, Safran H, Hoffman JP, Konski A, Benson AB, Macdonald JS, Kudrimoti MR, Fromm ML, Haddock MG, Schaefer P, Willett CG, Rich TA. Fluorouracil vs gemcitabine chemotherapy before and after fluorouracil-based chemoradiation following resection of pancreatic adenocarcinoma: a randomized controlled trial. JAMA. 2008 Mar 5;299(9):1019-26. doi: 10.1001/jama.299.9.1019. PMID 18319412
- [Background] Hattangadi et al Cancer 8/15/2009 p 3640-3650
- [Background] Nichols RC Jr, Huh SN, Prado KL, Yi BY, Sharma NK, Ho MW, Hoppe BS, Mendenhall NP, Li Z, Regine WF. Protons offer reduced normal-tissue exposure for patients receiving postoperative radiotherapy for resected pancreatic head cancer. Int J Radiat Oncol Biol Phys. 2012 May 1;83(1):158-63. doi: 10.1016/j.ijrobp.2011.05.045. Epub 2012 Jan 13. PMID 22245197
- [Background] Kalser MH, Ellenberg SS. Pancreatic cancer. Adjuvant combined radiation and chemotherapy following curative resection. Arch Surg. 1985 Aug;120(8):899-903. doi: 10.1001/archsurg.1985.01390320023003. PMID 4015380
- [Background] Klinkenbijl JH, Jeekel J, Sahmoud T, van Pel R, Couvreur ML, Veenhof CH, Arnaud JP, Gonzalez DG, de Wit LT, Hennipman A, Wils J. Adjuvant radiotherapy and 5-fluorouracil after curative resection of cancer of the pancreas and periampullary region: phase III trial of the EORTC gastrointestinal tract cancer cooperative group. Ann Surg. 1999 Dec;230(6):776-82; discussion 782-4. doi: 10.1097/00000658-199912000-00006. PMID 10615932
- [Background] Van Laethem JL, Van Cutsem E, Hammel P, Mornex F, Azria D, Van Tienhoven G, Peeters M, Praet M, Budach V, Haustermans K et al. Adjuvant chemotherapy alone vs. chemoradiation after curative resection for pancreatic cancer: phase II/III trial of the EORTC/FFCD/GERCOR groups.